CLINICAL TRIAL: NCT00357123
Title: Use of Rosuvastatin in Integral Management of Abdominal Sepsis
Brief Title: Effect of Rosuvastatin in Abdominal Sepsis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: UASLP, Martin Sanchez Aguilar
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 28-08 ROAS
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2010-09

CONDITIONS: Sepsis
Keywords: abdominal sepsis; sepsis; rosuvastatin
MeSH Terms: conditions — Sepsis; Intraabdominal Infections | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg 10 days daily since abdominal sepsis diagnosis
  Other Names: Crestor

SUMMARY:
The purpose of this study is to determine whether rosuvastatin is effective as a coadjuvant drug in the integral management of abdominal sepsis acknowledged by surgery.

DETAILED DESCRIPTION:
The sepsis is often lethal, the mortality's ranks are identified among 25 to 70%, this depends on definition, severity and co-morbidities. The number of deaths by sepsis could be similar to myocardial infarct. Patients who get shock have 26-fold risk of death.

In preliminary studies have been observed, that patients with treatment with statin have minor incidence of severe sepsis. A retrospective study suggests the association between using statins and reduction of bacteriemia by Gram negatives and S. aureus.

There are many experimental studies which demonstrate the possible profit in sepsis. However there are no clinical prospective studies for determinate if statins are effective in management of sepsis. The investigators designed this study to demonstrate the utility of rosuvastatin in one kind of sepsis, abdominal sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Man or women > 18 and < 80 years old with abdominal sepsis, confirmed diagnosis by surgery of broad peritonitis before 48 hours in progression
2. Injury by steel or firearm with contaminated abdominal cavity
3. APACHE II major or equal than 8
4. Acceptance to be included

Exclusion Criteria:

1. Ingestion of: fibrates, niacin, cyclosporin, azoles, macrolides, inhibitors of protease, nefazodone, verapamil, diltiazem, amiodarone
2. Hypovolemic shock III and IV after get surgery
3. Cardio-respiratory failure pre or trans surgery
4. Allergy to used drug
5. Use previous of statin
6. Hepatopathy or myopathy and(or) history, hepatic failure (Child B y C)
7. Management in other Hospital
8. Pregnancy
9. Thoracic injury, head injury (moderate and severe), multiple fractures or with bone exposition, rectal injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Plasmatic levels of Interleukine 6 and 1B, and Tumor Necrosis Factor alpha (pg/dL) | day 3

SECONDARY OUTCOMES:
Number of survivors | 1 week after randomization
  in-patient follow-up will be considered as well
Plasmatic levels of Reactive C Protein (mg/dL) | day 3
Classification of severity by APACHE II scale | day 3
Incidence of complications or secondary effects | day 1, 3, 7, 14 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sanchez-Aguilar, MSc, Principal Investigator — Experimental Surgery , Universidad Autonoma de San Luis Potosi
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico